CLINICAL TRIAL: NCT02601417
Title: The Necessity of Bile Cultures in Patients With Acute Cholangitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Sang Hyub Lee, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015-1452
Record Dates: First submitted 2015-08-27; First posted 2015-11-10 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Acute Cholangitis
Keywords: Cholangitis; Bile culture; percutaneous transhepatic biliary drainage
MeSH Terms: conditions — Cholangitis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotics change is based on both blood and bile cultures (No Intervention): Empirical antibiotic therapy was initially conducted for patients. In the control group, the initial antibiotic regimen was maintained if both blood and bile cultures were negative or if all identified organisms were sensitive to empirical treatment. However, the empirical antibiotics were switched to appropriate antibiotics considering the results from blood and bile cultures if any organism demonstrated resistance.
  Following antibiotic modification in the experimental and control groups, additional biliary drainage procedures (ERCP or PTBD) were performed for considering ineffective drainage on the discretion of physicians.
- Antibiotics change is based only on the blood culture (Experimental): Empirical antibiotic therapy was initially conducted for patients. In experimental group, the antibiotic therapy was modified based only on the blood culture findings, where the blood cultures revealed insensitive organisms with the resistance to empirical antibiotics. The bile specimens from these patients were also obtained and cultured, but their results were not considered in the decision-making for antibiotic selection in the experimental group.
  Following antibiotic modification in the experimental and control groups, additional biliary drainage procedures (ERCP or PTBD) were performed for considering ineffective drainage on the discretion of physicians.
  Interventions: Other: Ignoring result of bile culture

INTERVENTIONS:
Other: Ignoring result of bile culture — the antibiotic therapy was modified based only on the blood culture findings, where the blood cultures revealed insensitive organisms with the resistance to empirical antibiotics. The bile specimens from these patients were also obtained and cultured, but their results were not considered in the decision-making for antibiotic selection in the experimental group
  Arms: Antibiotics change is based only on the blood culture

SUMMARY:
Acute cholangitis with obstructive jaundice is a condition which needs biliary drainage and appropriate antibiotics. Bile culture is an optional laboratory test according to 2013, 2018 Tokyo guideline, but the clinical significance is yet unproven. And its results might indicate less information of the true pathogen regarding normal flora. Previous study conducted at our institute found drug-resistant pathogens identified in bile culture had no impact on the outcome. So the investigators are conducting a multicenter randomized controlled trial comparing groups which considers both blood and bile culture as control and which considers only blood culture as trial group in order to prove bile culture provides no additional helpful clinical information.

DETAILED DESCRIPTION:
The investigators conducted a nationwide, prospective, multicenter, subject blinded, noninferiority RCT. Patients with acute cholangitis who met the specific inclusion criteria were enrolled. All the participants underwent a percutaneous transhepatic biliary drainage (PTBD) procedure to provide adequate drainage, and both bile and blood cultures were collected. A culture study was performed after obtaining the initial bile from the bile duct assessment during PTBD insertion. In this study, the patients who were conducted endoscopic retrograde cholangiopancreatography (ERCP) and biliary drainage were excluded to avoid unintended contamination by normal flora of gastrointestinal tract.

Initially, empirical broad-spectrum antibiotics, including metronidazole combined with third-generation cephalosporins or quinolones were administered for treating acute cholangitis. All participants provided informed consent after explaining the study details. Participants who consented to participate were then randomized.

The investigators recruited patients aged ≥20 years with suspected or confirmed acute cholangitis according to the 2013 and 2018 Tokyo guidelines. The exclusion criteria were (1) inability to provide informed consent, (2) no evidence of acute cholangitis diagnostics as per the guidelines, (3) development of organ failure before random allocation or organ failure by non-cholangitis causes, (4) undergoing bile culture tests after the onset of organ failure, (5) failure to have bile or blood culture tests, (6) patients who were already administered antibiotics for other conditions, (7) unsuccessful PTBD insertion, and (8) failure to achieve complete bile drainage via PTBD.

Empirical antibiotic therapy was initially conducted for both groups of patients. In the control group, the initial antibiotic regimen was maintained if both blood and bile cultures were negative or if all identified organisms were sensitive to empirical treatment. However, the empirical antibiotics were switched to appropriate antibiotics considering the results from blood and bile cultures if any organism demonstrated resistance. In experimental group, the antibiotic therapy was modified based only on the blood culture findings, where the blood cultures revealed insensitive organisms with the resistance to empirical antibiotics. The bile specimens from these patients were also obtained and cultured, but their results were not considered in the decision-making for antibiotic selection in the experimental group.

Following antibiotic modification in the experimental and control groups, additional biliary drainage procedures (ERCP or PTBD) were performed for considering ineffective drainage on the discretion of physicians.

The investigators carried out a per-protocol analysis that excluded patients who had received antibiotics prior to PTBD, which could have altered the microbial profile, those with lethal adverse events before the confirmation of blood or bile culture results, and those who had been administered changed antibiotics for infectious diseases other than acute cholangitis.

Student's t-test was used to analyze continuous variables with normal distribution, Mann-Whitney U-test was performed otherwise. Categorical variables were assessed with the chi-square test or Fisher's exact test. A p-value of ≤0.05 indicated significant differences, and the respective variables were regarded as covariates for adjustment in each analysis. Student's t-test and Mann-Whitney U-test were used to compare mortality and hospital stay duration. All the tests were two-sided, and a p-value of <0.05 was regarded as statistically significant. In the analyses of binary outcomes, the results are presented as point estimates for the between-group differences in the proportion of patients. The two-sided 95% confidence interval (CI) for these differences was calculated using the Wald method.

ELIGIBILITY:
The inclusion criteria

(1) patients aged ≥20 years with suspected or confirmed acute cholangitis according to the 2013 and 2018 Tokyo guidelines

The exclusion criteria

1. inability to provide informed consent
2. no evidence of acute cholangitis diagnostics as per the guidelines
3. development of organ failure before random allocation or organ failure by non-cholangitis causes
4. undergoing bile culture tests after the onset of organ failure
5. failure to have bile or blood culture tests
6. patients who were already administered antibiotics for other conditions
7. unsuccessful PTBD insertion
8. failure to achieve complete bile drainage via PTBD

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Estimated)
Dates: Start 2015-08-27 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Organ Failure | during hospitalization and empirical antibiotic administration. (From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months)
  Shock, AKI, altered mentality, Acute respiratory distress

SECONDARY OUTCOMES:
Hospital days | through study completion, an average of 1 month
  The duration of hospital stay covered the period from randomization to discharge for the management of acute cholangitis
Re-intervention for biliary drainage | through study completion, an average of 1 month
  The frequency of reintervention for biliary drainage was the proportion of patients undergoing additional procedures during the study period.
Mortality | through study completion, an average of 1 month
  Mortality rate was the proportion of patients experiencing death during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hyub Lee, MD. PhD., Principal Investigator — Department of internal medicine and liver research institute, Seoul national university hospital, Seoul, Korea
Locations (1):
- Seoul National University Hospital, Seoul, South Korea